CLINICAL TRIAL: NCT06534489
Title: Surgical Strategy of NSCLC Patients After Neo-adjuvant or Induction Treatment
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Huadong Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: RTS-021
Record Dates: First submitted 2024-05-22; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-05

CONDITIONS: Non-small Cell Lung Cancer; Surgery
Keywords: lung cancer; Neo-adjuvant treatment; pneumonectomy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolled patients: After the patients were enrolled in the group, further relevant examinations (chest enhancement CT, PET-CT (optional), cranial MR, bronchoscopy, cardiac ultrasound, pulmonary function, electrocardiogram, blood tests) were completed, contraindications to surgery were ruled out, and the patients were evaluated to receive neo-adjuvant immuno-chemotherapy. After treatment, patients should be re-evaluated and amenable to surgical treatment after multidisciplinary discussion (thoracic surgery, respiratory medicine, radiology), and open or minimally invasive radical lung cancer surgery and systematic lymph node dissection were performed, including pneumonectomy, lobectomy, double lobectomy, extended lobectomy or sleeve lobectomy. The perioperative complications, lymph node dissection, R0 clearance rate, 3-year event-free survival rate, overall and disease-free survival rate, quality of life, and pulmonary function were recorded and evaluated.
  Interventions: Procedure: neoadjuvant immuno-chemotherapy and surgery

INTERVENTIONS:
Procedure: neoadjuvant immuno-chemotherapy and surgery — After enrolled, patients should receive neo-adjuvant immuno-chemotherapy and a re-evaluation will be performed after treatment to decide surgery strategy.

SUMMARY:
Lung cancer is one of the most common malignant tumors worldwide and has the highest mortality rate among malignant tumors. In recent years, with the gradual development of therapeutic modalities such as targeted therapy and immunotherapy, the overall survival of lung cancer patients has improved significantly. However, late tumor staging at the time of diagnosis often leaves patients with only pneumonectomy, which affects the prognosis with a higher rate of postoperative complications than lobectomy, poorer quality of life and the possible loss of the opportunity to continue adjuvant therapy. Our group proposes to conduct this single-arm prospective clinical study to investigate the feasibility, safety and prognosis of the conversion from pneumonectomy to lobectomy after neoadjuvant or induction therapy in patients with operable non-small cell lung cancer.

DETAILED DESCRIPTION:
We propose to conduct a multicenter, single-arm prospective clinical study to investigate the feasibility, safety and prognosis of the conversion from pneumonectomy to lobectomy after neoadjuvant or induction therapy in patients with operable non-small cell lung cancer. The anticipated sample size is 50 patients. Study will last 5 years.

After the patients were enrolled in the group, further relevant examinations (chest enhancement CT, PET-CT (optional), cranial MR, bronchoscopy, cardiac ultrasound, pulmonary function, electrocardiogram, blood tests) were completed, contraindications to surgery were ruled out, and the patients were evaluated to receive neoadjuvant or induction chemo-immunotherapy after multidisciplinary discussion (thoracic surgery, respiratory medicine, radiology). After the patients completed these treatments, systemic preoperative examinations should be underwent (chest enhancement CT, PET-CT (optional), cranial MR, bronchoscopy, cardiac ultrasound, pulmonary function, electrocardiogram, blood tests) and open or minimally invasive radical lung cancer surgery and systematic lymph node dissection were performed. The perioperative complications, lymph node dissection, R0 clearance rate, 3-year event-free survival rate, overall and disease-free survival rate, quality of life, and pulmonary function were recorded and evaluated.

The surgical strategies include pneumonectomy, double lobectomy, sleeve lobectomy and lobectomy.

The patients will be followed up in one and three months after surgery. Then every three months in first year, every six months after one year of operation, with blood routine, biochemistry, tumor indexes, and chest CT examination at each visit. Within one year after surgery, head MR was performed every six months and PET-CT was performed at one year, and after one year after surgery, head MR was performed every six months and PET-CT was performed every year.

The researchers will contact the study participants or their families via the Internet or telephone to inform them of the treatment schedule and remind them of follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* The patients voluntarily participate in the study, have good compliance, can cooperate with the requirements of the experiment to complete the observation and follow-up, and sign the informed consent form.
* Aged over 18 years old, under 75 years old; male and female are not limited;
* Pathologically confirmed non-small cell lung cancer with clinical stage T2-4N0-2, resectable non-small cell lung cancer, potentially needing pneumonectomy and receiving neoadjuvant or induction therapy.
* ASA score: Grade I-III;
* The cardiopulmonary function evaluation can meet the requirements for radical lung cancer surgery, and the liver and kidney functions are normal.

Exclusion Criteria:

* Those with serious cardiac, pulmonary, hepatic, and renal dysfunctions, unable to tolerate the surgery;
* Those with uncontrollable neurological or psychiatric diseases or mental disorders, poor compliance, and being unable to cooperate and describe the treatment response.
* Those who are going to undergo emergency surgery or palliative surgery due to lung abscess or hemoptysis.
* Those who have been treated, or are undergoing neoadjuvant or induction radiotherapy or targeted therapy.
* Those who have a combined history of other malignant tumors
* Those who have a history of thoracic surgery
* Those who are pregnant or breastfeeding women
* Patients of childbearing age who refuse to use contraception.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Source of study subjects: outpatients Recruitment location: Thoracic Surgery and Respiratory Medicine Clinic of participant centers.
  Recruitment method:Through WeChat public number, departmental website and other online channels to publish recruitment information.
  The researchers conducted a study on the lungs of patients attending outpatient clinics. After preliminary evaluation of lung cancer patients in the outpatient clinic of Ruijin Hospital and identification of those who are potentially eligible for enrollment, as well as improvement of chest CT, PET-CT（optional）, cardiac ultrasound, lung function and other auxiliary examinations, and after it is clear that they are eligible for enrollment, subjects will be informed of the study and will sign an informed consent form.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-08-31 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Tumor R0 resection rate (lobectomy) | Two weeks after surgery according to Frozen pathologic test and Paraffin pathologic test
  the proportion of patients with complete tumor removal by lobectomy, as evaluated by the pathologic findings of postoperative lung cancer specimens

SECONDARY OUTCOMES:
Lymph node dissection | Two weeks after surgery according to Paraffin pathologic test
  Record the total number of lymph node dissection, the number of stations of lymph node dissection, and the number of lymph node dissection at each station during the operation,and evaluate them according to the pathologic results.
Duration of surgery | 1 month after surgery
  Record the duration of surgery in minute（min），evaluated by surgical records and perioperative clinical manifestations, laboratory tests, physical examination
Intraoperative bleeding | 1 month after surgery
  Record intraoperative bleeding in milliliter （ml）, evaluated by surgical records and perioperative clinical manifestations, laboratory tests, physical examination
Incidence of intraoperative accidents | 1 month after surgery
  Record the incidence of intraoperative accidents in rate（%）, including bleeding，injury to normal tissue or organ， evaluated by surgical records and perioperative clinical manifestations, laboratory tests, physical examination
Postoperative short-term efficacy indicators | 1 month after surgery
  record the length of postoperative hospitalization (days), survival within 30 days after surgery, and evaluate through postoperative follow-up
Perioperative complication rate | 1 month after surgery
  Evaluated by clinical manifestations, laboratory tests, and physical examination
3-year disease-free survival rate | When all enrolled patients complete 3-year follow-up
  defined as the proportion of patients without tumor recurrence or metastasis 3 years after surgery, evaluated by postoperative follow-up
3-year overall survival rate | When all enrolled patients complete 3-year follow-up
  defined as the proportion of patients who are still alive 3 years after surgery, and evaluated by postoperative follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin hospital, Shanghai, China

REFERENCES:
- [Background] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Akinyemiju TF, Al Lami FH, Alam T, Alizadeh-Navaei R, Allen C, Alsharif U, Alvis-Guzman N, Amini E, Anderson BO, Aremu O, Artaman A, Asgedom SW, Assadi R, Atey TM, Avila-Burgos L, Awasthi A, Ba Saleem HO, Barac A, Bennett JR, Bensenor IM, Bhakta N, Brenner H, Cahuana-Hurtado L, Castaneda-Orjuela CA, Catala-Lopez F, Choi JJ, Christopher DJ, Chung SC, Curado MP, Dandona L, Dandona R, das Neves J, Dey S, Dharmaratne SD, Doku DT, Driscoll TR, Dubey M, Ebrahimi H, Edessa D, El-Khatib Z, Endries AY, Fischer F, Force LM, Foreman KJ, Gebrehiwot SW, Gopalani SV, Grosso G, Gupta R, Gyawali B, Hamadeh RR, Hamidi S, Harvey J, Hassen HY, Hay RJ, Hay SI, Heibati B, Hiluf MK, Horita N, Hosgood HD, Ilesanmi OS, Innos K, Islami F, Jakovljevic MB, Johnson SC, Jonas JB, Kasaeian A, Kassa TD, Khader YS, Khan EA, Khan G, Khang YH, Khosravi MH, Khubchandani J, Kopec JA, Kumar GA, Kutz M, Lad DP, Lafranconi A, Lan Q, Legesse Y, Leigh J, Linn S, Lunevicius R, Majeed A, Malekzadeh R, Malta DC, Mantovani LG, McMahon BJ, Meier T, Melaku YA, Melku M, Memiah P, Mendoza W, Meretoja TJ, Mezgebe HB, Miller TR, Mohammed S, Mokdad AH, Moosazadeh M, Moraga P, Mousavi SM, Nangia V, Nguyen CT, Nong VM, Ogbo FA, Olagunju AT, Pa M, Park EK, Patel T, Pereira DM, Pishgar F, Postma MJ, Pourmalek F, Qorbani M, Rafay A, Rawaf S, Rawaf DL, Roshandel G, Safiri S, Salimzadeh H, Sanabria JR, Santric Milicevic MM, Sartorius B, Satpathy M, Sepanlou SG, Shackelford KA, Shaikh MA, Sharif-Alhoseini M, She J, Shin MJ, Shiue I, Shrime MG, Sinke AH, Sisay M, Sligar A, Sufiyan MB, Sykes BL, Tabares-Seisdedos R, Tessema GA, Topor-Madry R, Tran TT, Tran BX, Ukwaja KN, Vlassov VV, Vollset SE, Weiderpass E, Williams HC, Yimer NB, Yonemoto N, Younis MZ, Murray CJL, Naghavi M. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-Years for 29 Cancer Groups, 1990 to 2016: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2018 Nov 1;4(11):1553-1568. doi: 10.1001/jamaoncol.2018.2706. PMID 29860482
- [Background] Saji H, Okada M, Tsuboi M, Nakajima R, Suzuki K, Aokage K, Aoki T, Okami J, Yoshino I, Ito H, Okumura N, Yamaguchi M, Ikeda N, Wakabayashi M, Nakamura K, Fukuda H, Nakamura S, Mitsudomi T, Watanabe SI, Asamura H; West Japan Oncology Group and Japan Clinical Oncology Group. Segmentectomy versus lobectomy in small-sized peripheral non-small-cell lung cancer (JCOG0802/WJOG4607L): a multicentre, open-label, phase 3, randomised, controlled, non-inferiority trial. Lancet. 2022 Apr 23;399(10335):1607-1617. doi: 10.1016/S0140-6736(21)02333-3. PMID 35461558
- [Background] Altorki N, Wang X, Kozono D, Watt C, Landrenau R, Wigle D, Port J, Jones DR, Conti M, Ashrafi AS, Liberman M, Yasufuku K, Yang S, Mitchell JD, Pass H, Keenan R, Bauer T, Miller D, Kohman LJ, Stinchcombe TE, Vokes E. Lobar or Sublobar Resection for Peripheral Stage IA Non-Small-Cell Lung Cancer. N Engl J Med. 2023 Feb 9;388(6):489-498. doi: 10.1056/NEJMoa2212083. PMID 36780674
- [Background] Jones GD, Tan KS, Caso R, Dycoco J, Park BJ, Bott MJ, Molena D, Huang J, Isbell JM, Bains MS, Jones DR, Rocco G. Time-varying analysis of readmission and mortality during the first year after pneumonectomy. J Thorac Cardiovasc Surg. 2020 Jul;160(1):247-255.e5. doi: 10.1016/j.jtcvs.2020.02.086. Epub 2020 Mar 7. PMID 32249082
- [Background] Shapiro M, Swanson SJ, Wright CD, Chin C, Sheng S, Wisnivesky J, Weiser TS. Predictors of major morbidity and mortality after pneumonectomy utilizing the Society for Thoracic Surgeons General Thoracic Surgery Database. Ann Thorac Surg. 2010 Sep;90(3):927-34; discussion 934-5. doi: 10.1016/j.athoracsur.2010.05.041. PMID 20732520
- [Background] Yang J, Xia Y, Yang Y, Ni ZZ, He WX, Wang HF, Xu XX, Yang YL, Fei K, Jiang GN. Risk factors for major adverse events of video-assisted thoracic surgery lobectomy for lung cancer. Int J Med Sci. 2014 Jun 11;11(9):863-9. doi: 10.7150/ijms.8912. eCollection 2014. PMID 25013365
- [Background] Kozower BD, Sheng S, O'Brien SM, Liptay MJ, Lau CL, Jones DR, Shahian DM, Wright CD. STS database risk models: predictors of mortality and major morbidity for lung cancer resection. Ann Thorac Surg. 2010 Sep;90(3):875-81; discussion 881-3. doi: 10.1016/j.athoracsur.2010.03.115. PMID 20732512
- [Background] Pricopi C, Mordant P, Rivera C, Arame A, Foucault C, Dujon A, Le Pimpec Barthes F, Riquet M. Postoperative morbidity and mortality after pneumonectomy: a 30-year experience of 2064 consecutive patients. Interact Cardiovasc Thorac Surg. 2015 Mar;20(3):316-21. doi: 10.1093/icvts/ivu417. Epub 2014 Dec 8. PMID 25487232
- [Background] Schneider L, Farrokhyar F, Schieman C, Shargall Y, D'Souza J, Camposilvan I, Hanna WC, Finley CJ. Pneumonectomy: the burden of death after discharge and predictors of surgical mortality. Ann Thorac Surg. 2014 Dec;98(6):1976-81; discussion 1981-2. doi: 10.1016/j.athoracsur.2014.06.068. Epub 2014 Oct 3. PMID 25282164
- [Background] Kim AW, Boffa DJ, Wang Z, Detterbeck FC. An analysis, systematic review, and meta-analysis of the perioperative mortality after neoadjuvant therapy and pneumonectomy for non-small cell lung cancer. J Thorac Cardiovasc Surg. 2012 Jan;143(1):55-63. doi: 10.1016/j.jtcvs.2011.09.002. Epub 2011 Nov 4. PMID 22056364
- [Background] Jones GD, Caso R, Tan KS, Dycoco J, Adusumilli PS, Bains MS, Downey RJ, Huang J, Isbell JM, Molena D, Park BJ, Rocco G, Rusch VW, Sihag S, Jones DR, Bott MJ. Propensity-matched Analysis Demonstrates Long-term Risk of Respiratory and Cardiac Mortality After Pneumonectomy Compared With Lobectomy for Lung Cancer. Ann Surg. 2022 Apr 1;275(4):793-799. doi: 10.1097/SLA.0000000000004065. PMID 32541218
- [Background] Riquet M, Mordant P, Pricopi C, Legras A, Foucault C, Dujon A, Arame A, Le Pimpec-Barthes F. A review of 250 ten-year survivors after pneumonectomy for non-small-cell lung cancer. Eur J Cardiothorac Surg. 2014 May;45(5):876-81. doi: 10.1093/ejcts/ezt494. Epub 2013 Oct 16. PMID 24132299
- [Background] Sartipy U. Prospective population-based study comparing quality of life after pneumonectomy and lobectomy. Eur J Cardiothorac Surg. 2009 Dec;36(6):1069-74. doi: 10.1016/j.ejcts.2009.05.011. Epub 2009 Jul 5. PMID 19581107
- [Background] Balduyck B, Hendriks J, Lauwers P, Van Schil P. Quality of life after lung cancer surgery: a prospective pilot study comparing bronchial sleeve lobectomy with pneumonectomy. J Thorac Oncol. 2008 Jun;3(6):604-8. doi: 10.1097/JTO.0b013e318170fca4. PMID 18520798
- [Background] Lococo F, Sassorossi C, Nachira D, Chiappetta M, Petracca Ciavarella L, Vita E, Boldrini L, Evangelista J, Cesario A, Bria E, Margaritora S. Prognostic Factors and Long-Term Survival in Locally Advanced NSCLC with Pathological Complete Response after Surgical Resection Following Neoadjuvant Therapy. Cancers (Basel). 2020 Nov 30;12(12):3572. doi: 10.3390/cancers12123572. PMID 33265905
- [Background] Arriagada R, Bergman B, Dunant A, Le Chevalier T, Pignon JP, Vansteenkiste J; International Adjuvant Lung Cancer Trial Collaborative Group. Cisplatin-based adjuvant chemotherapy in patients with completely resected non-small-cell lung cancer. N Engl J Med. 2004 Jan 22;350(4):351-60. doi: 10.1056/NEJMoa031644. PMID 14736927
- [Background] Forde PM, Spicer J, Lu S, Provencio M, Mitsudomi T, Awad MM, Felip E, Broderick SR, Brahmer JR, Swanson SJ, Kerr K, Wang C, Ciuleanu TE, Saylors GB, Tanaka F, Ito H, Chen KN, Liberman M, Vokes EE, Taube JM, Dorange C, Cai J, Fiore J, Jarkowski A, Balli D, Sausen M, Pandya D, Calvet CY, Girard N; CheckMate 816 Investigators. Neoadjuvant Nivolumab plus Chemotherapy in Resectable Lung Cancer. N Engl J Med. 2022 May 26;386(21):1973-1985. doi: 10.1056/NEJMoa2202170. Epub 2022 Apr 11. PMID 35403841

DOCUMENTS (2):
  • Study Protocol (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT06534489/Prot_000.pdf
  • Informed Consent Form (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT06534489/ICF_001.pdf